CLINICAL TRIAL: NCT00914966
Title: A Phase 4 Study to Evaluate the Safety and Effect of Escalating Doses of CINRYZE® (C1 Inhibitor [Human]) as Prophylactic Therapy in Subjects With Inadequately Controlled Hereditary Angioedema Attacks
Brief Title: A Study to Evaluate the Safety and Effect of Escalating Doses of CINRYZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0624-400; SHP616-400 (Other: Sponsor)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; SERPING1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CINRYZE (Experimental): There were 3 potential dose escalation steps:
  * Step 1: 1500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks
  * Step 2: 2000 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks
  * Step 3: 2500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks
  Interventions: Biological: C1 inhibitor (human) [C1 INH]

INTERVENTIONS:
Biological: C1 inhibitor (human) [C1 INH]
  Other Names: CINRYZE; C1 esterase inhibitor (human)

SUMMARY:
The objectives of the study were:

1. To assess the safety and tolerability of escalating doses of CINRYZE.
2. To assess the effect of an escalating dose algorithm for CINRYZE on hereditary angioedema (HAE) attack rates.
3. To assess the immunogenicity of CINRYZE.

DETAILED DESCRIPTION:
Qualifying subjects entered a 3-step dose escalation algorithm:

* Step 1: 1500 Units twice per week (starting dosing regimen for all subjects in the study)
* Step 2: 2000 Units twice per week
* Step 3: 2500 Units twice per week

Each step consisted of 12 weeks of safety monitoring, followed by calculation of average monthly angioedema attack rate based on subject reports of angioedema symptoms (regardless of intensity) and actual duration of therapy for that step.

If a subject was deemed a "success" at a given step and the investigator and medical monitor determined that it was safe for the subject to continue on that dose, the subject entered a 3 month follow-up period at that dose level with continued safety monitoring. The subject could not re-enter the study for purposes of dose escalation during the follow-up period.

If a subject was not deemed a "success," the subject initiated the next highest step of the dose escalation algorithm provided that the investigator and medical monitor agreed that dose escalation was appropriate. If at the end of Step 3 (2500 Units), a subject was not deemed a "success," then the Week 12 visit represented study completion and the subject was referred to the physician who manages their HAE care.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this protocol, subjects must:

1. Be ≥6 years of age and ≥25 kg body weight.
2. Have a confirmed diagnosis of HAE with a documented history of swelling of the face, extremities, gastrointestinal tract, genitalia, or larynx and a history of at least one of the following:

   * C1 INH gene mutation
   * C4 level below the lower limit of the reference range
   * C1 INH antigen level below the lower limit of the reference range
   * Functional C1 INH level below the lower limit of the reference range
   * Family history of HAE (i.e., grandparent, parent, sibling)
3. Have a history of >1.0 HAE attack per month (average) of any severity during the 3 consecutive months prior to screening while receiving the recommended CINRYZE dosing of 1000 Units every 3 to 4 days via intravenous injection.
4. If an adult, be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.

   OR
5. If a child, have a parent/legal guardian who is willing and able to provide written informed consent for the child to participate in the study (with assent from the child when appropriate).

Exclusion Criteria:

To be eligible for this protocol, subjects must not:

1. Have, as determined by the investigator and/or the sponsor's medical monitor, any surgical or medical condition that could interfere with the administration of study drug or interpretation of study results.
2. Have a history of abnormal blood clotting or other coagulopathy.
3. Be taking prescription anticoagulant medication.
4. Have a history of allergic reaction to CINRYZE or other blood products.
5. Have participated in any other investigational drug study within the past 30 days (other than CINRYZE protocols).
6. Have received any blood products (other than CINRYZE) within 60 days prior to screening.
7. Have any of the following laboratory values at screening:

   * Hemoglobin <8 g/dL
   * White blood cell count <2 x 10^9/L or >20 x 10^9/L
   * Platelet count <50 x 10^9/L or >400 x 10^9/L
   * Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.0 x the upper limit of normal
   * Blood urea nitrogen and/or creatinine >2.0 x the upper limit of normal
8. Be pregnant or breastfeeding.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2012-05-24 (Actual); Study Completion 2012-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (11):
  - Allergy, Asthma and Immunology Associates, Scottsdale, Arizona
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Winthrop University Hospital, Mineola, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - East Tennessee Center for Clinical Research, Knoxville, Tennessee
  - Bryan, Texas
  - AARA Research Center, Dallas, Texas
  - Marycliff Allergy Specialist, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- CINRYZE: There were 3 potential dose escalation steps: - Step 1: 1500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks (starting dosing regimen for all subjects in the study) - Step 2: 2000 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks - Step 3: 2500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks
Period: Step 1: 1500 Units
Arm/Group | CINRYZE
Started | 20
Completed | 18 (5/18 subjects completing Step 1 (1500 Units) entered the 3 month follow-up and did not dose escalate)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: Step 2: 2000 Units
Arm/Group | CINRYZE
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Step 3: 2500 Units
Arm/Group | CINRYZE
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CINRYZE
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (15.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events, Hospitalizations, Thrombotic Events, Treatment-emergent C1 INH Antibodies, Post-baseline Toxicity Grade Increases in Clinical Laboratory Parameters, and Post-dose Vital Signs Changes of Potential Clinical Importance
Description: Events reported during the 3 month follow-up period are counted with the dose level at which they occurred.
Time Frame: 12 to 24 weeks at each dose level
Measure: Number; unit: participants
Groups:
- Step 1: 1500 Units: 1500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks.
- Step 2: 2000 Units: 2000 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks.
- Step 3: 2500 Units: 2500 Units of CINRYZE (C1 inhibitor [human]) administered by IV infusion twice per week for 12 weeks.
Arm/Group | Step 1: 1500 Units | Step 2: 2000 Units | Step 3: 2500 Units
Number analyzed (Participants) | 20 | 13 | 12
participants
  Adverse events | 15 | 11 | 11
  Hospitalizations | 0 | 1 | 0
  Systemic thrombotic events | 0 | 0 | 0
  Local/catheter-related thrombotic events | 1 | 0 | 0
  Treatment-emergent C1 INH antibodies | 0 | 0 | 1
  Toxicity grade increases in laboratory parameters | 6 | 2 | 3
  Potential clinically important vital signs changes | 3 | 1 | 1

2. Secondary Outcome: Treatment Effect of Escalating Doses of CINRYZE on HAE Attack Rates
Description: Two definitions of success were applied in this study: 1) Per-protocol success - Average angioedema attack rate of ≤1.0 per month at the end of any dose escalation step (Week 12). The a priori definition of study success was 4 or more subjects with per-protocol success. 2) Investigator-determined success - Based on the investigator's clinical judgment, an average monthly angioedema attack rate demonstrating improvement sufficient for progression to follow-up. In addition, subjects who were not a per-protocol or investigator-determined success, but who experienced a reduction of >1.0 attack per month from their historical angioedema attack rate at the end of any dose escalation step (Week 12), were summarized.
Time Frame: 12 weeks at each dose level
Measure: Number; unit: participants
Arm/Group | Step 1: 1500 Units | Step 2: 2000 Units | Step 3: 2500 Units
Number analyzed (Participants) | 20 | 13 | 12
participants
  Per-protocol Success | 4 | 0 | 5
  Investigator-determined Success | 1 | 0 | 1
  Reduction of >1 attack/month from historical rate | 1 | 0 | 2
  Non-responder | 1 | 1 | 4

ADVERSE EVENTS:
Time Frame: 12 to 24 weeks at each dose level. Events reported during the 3 month follow-up period are counted with the dose level at which they occurred.
Arm/Group | Step 1: 1500 Units | Step 2: 2000 Units | Step 3: 2500 Units | All Subjects
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/13 | 1/12 | 2/20
Other Adverse Events (participants affected / at risk) | 12/20 | 5/13 | 6/12 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: 1500 Units (N=20) | Step 2: 2000 Units (N=13) | Step 3: 2500 Units (N=12) | All Subjects (N=20)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 — Not related to study drug
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 — Laryngeal HAE attack; Not related to study drug
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1 — Not related to study drug
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: 1500 Units (N=20) | Step 2: 2000 Units (N=13) | Step 3: 2500 Units (N=12) | All Subjects (N=20)
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 3 | 5 — 83% mild, 17% moderate
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 3 — 100% mild
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 2 — 100% mild
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 — 100% moderate
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 — 50% mild, 50% severe
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2 — 33% mild, 33% moderate, 33% severe
Medical device complication (General disorders) | 2 | 0 | 0 | 2 — 100% mild
Peripheral edema (General disorders) | 2 | 0 | 0 | 2 — 100% moderate
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 — 100% moderate
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 2 — 50% mild, 50% moderate
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 2 — 50% mild, 50% moderate
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 2 — 100% mild

LIMITATIONS AND CAVEATS:
Per Changes in the Planned Analyses:

The clinical presentation of disease manifestations and response to therapy are highly variable among patients with HAE and as such, the efficacy results from this study are presented in this report by individual participant in narrative summaries rather than as summary statistics.

Thus, one outcome measure (Use of rescue therapy and/or other therapy for treatment of HAE symptoms) is not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to Sponsor for pre-review. If Sponsor requests, PI must delete Sponsor confidential information before publication and/or delay publication for 60 days so Sponsor can file for patents or take other action to protect its patent rights.